CLINICAL TRIAL: NCT05533138
Title: Guided-internet Cognitive Behavioral Therapy for Antenatal Depression - Treatment Effects, Assessment Modalities and Extra Support.
Brief Title: Internet CBT for Antenatal Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Marie Bendix, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-06049
Record Dates: First submitted 2022-06-27; First posted 2022-09-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Antenatal Depression
Keywords: Cognitive behavior therapy; Internet treatment; Self-help treatment; Perinatal support
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Multiple Assignment Randomized Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded for allocation to perinatal extra support in addition to therapist-guided internet CBT treatment.
  Outcome is assessed by an independent assessor who is blind for whether patient chose or was allocated to assessment modality and whether patient received extra-support or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Assessment form allocated by chance & guided ICBT for antenatal depression (Active Comparator): Patients are randomized to assessment modality (telephone, video or face-to-face visit) of a perinatal psychiatric semi-structured assessment & and are randomised to treatment with internet-CBT for antenatal depression without extra-support (10 weeks)
  Interventions: Behavioral: Therapist Guided Internet-CBT for antenatal depression; Behavioral: Diagnostic assessment by telephone, video or face-to face - Allocation by chance
- Assessment form allocated by choice & guided ICBT for antenatal depression (Active Comparator): Patients choose assessment modality (telephone, video or face-to-face visit) of a perinatal psychiatric semi-structured assessment & are randomised to treatment with internet-CBT for antenatal depression without extra-support (10 weeks)
  Interventions: Behavioral: Therapist Guided Internet-CBT for antenatal depression; Behavioral: Diagnostic assessment by telephone, video or face-to face - Allocation by choice
- Assessment form allocated by chance & guided ICBT for antenatal depression with extra support (Experimental): Patients are randomized to assessment modality (telephone, video or face-to-face visit) of a perinatal psychiatric semi-structured assessment & and are randomised to treatment with internet-CBT for antenatal depression with extra-support
  Interventions: Behavioral: Therapist Guided Internet-CBT for antenatal depression and perinatal extra support.; Behavioral: Diagnostic assessment by telephone, video or face-to face - Allocation by chance
- Assessment form allocated by choice & guided ICBT for antenatal depression with extra support (Experimental): Patients choose assessment modality (telephone, video or face-to-face visit) of a perinatal psychiatric semi-structured assessment & are randomised to treatment with internet-CBT for antenatal depression with extra-support (10 weeks)
  Interventions: Behavioral: Therapist Guided Internet-CBT for antenatal depression and perinatal extra support.; Behavioral: Diagnostic assessment by telephone, video or face-to face - Allocation by choice

INTERVENTIONS:
Behavioral: Therapist Guided Internet-CBT for antenatal depression — A 10 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for depression adapted for antenatal depression.
  Arms: Assessment form allocated by chance & guided ICBT for antenatal depression; Assessment form allocated by choice & guided ICBT for antenatal depression
Behavioral: Therapist Guided Internet-CBT for antenatal depression and perinatal extra support. — A 10 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for depression adapted for antenatal depression. Additionally, up to three supportive contacts with a midwife or perinatal mental health nurse to support ICBT treatment and adress general pregnancy related health problems.
  Arms: Assessment form allocated by chance & guided ICBT for antenatal depression with extra support; Assessment form allocated by choice & guided ICBT for antenatal depression with extra support
Behavioral: Diagnostic assessment by telephone, video or face-to face - Allocation by chance — Structured diagnostic perinatal psychiatric assessment of women screening positive for antenatal depression (pregnancy week 8-29) by telephone, video or in a face-to-face meeting. Assessment form allocation by chance.
  Arms: Assessment form allocated by chance & guided ICBT for antenatal depression; Assessment form allocated by chance & guided ICBT for antenatal depression with extra support
Behavioral: Diagnostic assessment by telephone, video or face-to face - Allocation by choice — Structured diagnostic perinatal psychiatric assessment of women screening positive for antenatal depression (pregnancy week 8-29) by telephone, video or in a face-to-face meeting. Assessment form allocation based on patient preference.
  Arms: Assessment form allocated by choice & guided ICBT for antenatal depression; Assessment form allocated by choice & guided ICBT for antenatal depression with extra support

SUMMARY:
Pregnant women in pregnancy week 8-29 screening positive for antenatal depression will be randomized to either choose or to be allotted by chance to different forms of diagnostic assessment; i.e. telephone, video or face-to-face assessment.

Those diagnosed with mild to moderate major depression will then be randomized to treatment with therapist-guided Internet-delivered Cognitive Behavioral Therapy (ICBT) adapted for women suffering from antenatal depression or to the same treatment with addition of up to three contacts with extra support by a midwife or experienced perinatal mental health nurse.

The primary aim is to assess whether extrasupport in addition to internet-guided pregnancy adapted ICBT decreases depressive symptoms more than internet-guided pregnancy adapted ICBT only. Secondary aims include effects of extrasupport and assessment mode on treatment satisfaction, fidelity and credibility.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate major depression
* Pregnant at treatment start
* Regular contact with maternity mental health clinic
* > 18 years old
* Being able to start the treatment earliest in gestational week 8 and latest in gestational week 30
* Stable medication for depression and/or other psychiatric conditions for at least 3 weeks.
* Being able to participate in the treatment during the treatment time and having access to and being able to use the internet and mobile phone during the treatment time
* Being able to understand the Swedish language orally and in writing

Exclusion Criteria:

* Montgomery-Åsberg Depression Rating Scale-Self report version (MADRS-S) score below 15 (symptoms of depression to low) or above 35 (severe depression)
* High risk of self harm or suicide (based on semi-structured clinical suicide risk assessment)
* Psychiatric comorbidity, disability, somatic disorder, or pregnancy complications that prevent treatment participation or that can be negatively affected or compose a risk for the fetus by treatment participation
* Ongoing psychological treatment with similar content

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale, self-rating version (MADRS-S) | Baseline to post-treatment (10 weeks) and to 8-10 weeks post-partum
  A 9-item self-rated measure of depression severity that also screens for suicidality (Montgomery & Asberg, 1979). Scores range from 0 to 54 points with 13-19 points indicating mild depression, 20-34 points indicating moderate depression and 35-54 points indicating severe depression

SECONDARY OUTCOMES:
Change in Edinburgh Postnatal Depression Scale (EPDS) | Baseline to post-treatment (10 weeks) and to 8-10 weeks post-partum
  Self-rated measure of antenatal depression (Cox, Holden & Sagovsky, 1987) used for screening of perinatal depression and also as a severity measure. Scores range from 0 to 30 with 13 or more points being the cut off for depression during pregnancy. This scale is validated for Swedish pregnant women (Rubertsson et al., 2011).
Remission of major depression (DSM-5) | Post-treatment (10 weeks)
  Diagnostic assessment of major depression assessed by clinician in the same way as before treatment with the depression module of the SCID-I diagnostic interview based on DSM-5 (Spitzer et al., 1992).
Remission of major depression (DSM-5) | 8-10 weeks postpartum.
  Diagnostic assessment of major depression assessed by clinician in the same way as before treatment with the depression module of the SCID-I diagnostic interview based on DSM-5 (Spitzer et al., 1992).
Change in Generalized Anxiety Disorder-7 (GAD-7) | Screening to post-treatment (10 weeks) and to 8-10 weeks post-partum
  7-item self-assessment measure of symptoms of anxiety and worry (Spitzer et al., 2006). Scores range from 0 to 21 points with 10 points and above indicating clinical levels.
Change in self-rated Insomnia Severity Index (ISI) | Baseline to post-treatment (10 weeks) and to 8-10 weeks post-partum
  7-item, self-rated questionnaire measuring perceived severity of insomnia symptoms (Bastien, Vallières & Morin, 2001). Validated as an outcome measure for insomnia research. The scale includes seven items, scored on a 0-4 scale, that are summed to a range of 0-28. The score can be divided into four categories: no clinical insomnia (0-7), subthreshold insomnia (8-14), clinical insomnia of moderate severity (15-21) and severe clinical insomnia (22-28) (Sarsour et al., 2010).
Change in Work and Social Adjustment Scale (WSAS) | Baseline to post-treatment (10 weeks) and to 8-10 weeks post-partum
  Self-rated measure of level of impairment caused by a condition (Mundt et al. 2002). In this study two versions are used asking about impairment due to depression and due to pregnancy. Scores range from 0 to 40 with scores below 10 points indicating sub clinical impairment and scores above 20 indicating moderately severe impairment or worse.
Change in Euroqol (EQ-5D-5L) | Screening to post-treatment (10 weeks) and to 8-10 weeks post-partum
  Self-assessed, health related, quality of life questionnaire. 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (Hinz et al., 2014).
Change in Prenatal Attachment Inventory (PAI) | Screening to post-treatment (10 weeks)
  Self-rated measurement of attachment and mentalisation from the mother to the unborn child (Muller 1993; Pallant et al., 2014). 21-items scored on a 1-4 scale.
Change in Experience of close relationships (ENR) | Screening to 8-10 weeks post-partum
  Self-reported measurement of adult attachment style (Brennon et al., 1998; Fraley et al., 2000; Strand & Ståhl, 2008). 36 items scored on a 1-7 scale.
Change in Valentine Scale | Screening to 8-10 weeks post-partum
  7 item self-rated scale for measurement of satisfaction with the partner relationship (Burman et al., 2018). Range 0-21 with higher values indicating higher partner relationship satisfaction.
Change in Fear of birth scale (FOBS) | Screening to post-treatment (after 10 weeks) and to 8-10 weeks post-partum
  Self-assessment of fear and worry in relation to the approaching birth using two visual analogue scales (VAS)(Haines et al., 2015) with higher levels indicating increased fear and worry. Also used to assess fear and worry in relation to completed birth after delivery.
Change in Multidimensional Scale of Perceived Social Support (MSPSS) | Screening to 8-10 weeks post-partum
  Measures self-rated perceived social support (Zimet et al., 1988; Ekbäck et al., 2013). 12 items rated on a seven-point Likert-type response format (1 = very strongly disagree; 7 = very strongly agree). Range 12 to 84, with higher scores indicating higher perceived social support.
Change in Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Baseline to post-treatment (10 weeks) and to 8-10 weeks post-partum
  Measures healthcare consumption and productivity loss in patients with a psychiatric disorder (Bouwmans et al., 2013).
Change in Clinical Global Impression Severity Scale (CGI-S) | Post-assessment and post treatment (after week 10).
  7-item observer-rated scale that measures illness severity (CGI-S) (Guy 1976)
Change in Clinical Global clinical global improvement (CGI-I) | Post-assessment and post treatment (after week 10).
  7-item observer-rated scale that measures global improvement (CGI-I) (Guy 1976).

OTHER OUTCOMES:
Assessment of childbirth experience - The Childbirth experience scale (CEQ) | 8-10 weeks post-partum
  Measures the childbirth experience (Dencker et al., 2010) on a 22-item 4-point Likert scale assessing agreement with positive and negative statements ranging from 1 (Totally agree), 2 (Mostly agree), 3 (Mostly disagree) to 4 (Totally disagree).
Assessment of maternal bonding - Mother-to Infant-Bonding-Scale (S-MIBS) | 8-10 weeks post-partum
  Assesses maternal bonding with the infant during the postpartum period. Eight items ranging 0- 3 with higher values indicating more bonding challenges (Taylor et al. 2005, Morelius et al., 2020).
Assessment of Adverse events | Treatment week 2,4,6,8
  Patient rated adverse events.
Assessment of Adverse events | Post-treatment (10 weeks)
  Patient rated adverse events.
Assessment of Adverse events | 8-10 weeks post-partum
  Patient rated adverse events.
Assessment of Adverse events | Post-treatment (10 weeks).
  Clinician rated adverse events.
Assessment of treatment satisfaction - Client Satisfaction Questionnaire-8 (CSQ-8) | Post-treatment (10 weeks)
  Measures self-rated satisfaction with treatment with scores from 8 to 32 where 8-13 indicates poor, 14-19 fair, 20-25 good and 26-32 excellent satisfaction (Attkisson and Zwick, 1982; Smith et al. 2014)
Assessment of treatment satisfaction - Client Satisfaction Questionnaire-8 (CSQ-8) | 8-10 weeks postpartum
  Measures self-rated satisfaction with treatment with scores from 8 to 32 where 8-13 indicates poor, 14-19 fair, 20-25 good and 26-32 excellent satisfaction (Attkisson and Zwick, 1982; Smith et al. 2014)
Assessment of treatment credibility - Treatment Credibility Scale (TCS) | Treatment week 2
  The Treatment Credibility Scale is a version of the credibility/expectancy questionnaire (Devilly and Borkovec, 2000) assessing how well the respondent thinks the treatment would work for similar problems. Scores range from 5 to 50.
Assessment of treatment credibility - Treatment Credibility Scale (TCS) | Treatment week 4
  The Treatment Credibility Scale is a version of the credibility/expectancy questionnaire (Devilly and Borkovec, 2000) assessing how well the respondent thinks the treatment would work for similar problems. Scores range from 5 to 50.
Assessment of treatment fidelity | Post-treatment (10 weeks)
  Clinician rated structured assessment with instrument developed at the clinic for internet psychiatry.
Assessment of maternity health care, birth- and child related health and care outcomes - Swedish pregnancy and medical birth registers. | Pregnancy to 8-10 weeks postpartum
  Register data from the Swedish pregnancy and Medical Birth registers regering data on demographic, material health care, delivery care and child related outcomes will be linked by means of the unique personal identification number.
Assessment of empowerment | Post-assessment, post treatment (after week 10) and 8-10 weeks postpartum
  Patient rated empowerment rated with the 28-item "Empowerment Scale" (Rogers et al. 1997).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bendix, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Psychiatry Southwest, Department of CL Psychiatry & Internetpsychiatry, Stockholm, Sweden

REFERENCES:
- [Background] Forsell E, Bendix M, Hollandare F, Szymanska von Schultz B, Nasiell J, Blomdahl-Wetterholm M, Eriksson C, Kvarned S, Lindau van der Linden J, Soderberg E, Jokinen J, Wide K, Kaldo V. Internet delivered cognitive behavior therapy for antenatal depression: A randomised controlled trial. J Affect Disord. 2017 Oct 15;221:56-64. doi: 10.1016/j.jad.2017.06.013. Epub 2017 Jun 13. PMID 28628768
- See also: The homepage for the study where patients can register — https://dana.ki.se